CLINICAL TRIAL: NCT02049047
Title: Phase II Study of Everolimus in Patients With Thymoma and Thymic Carcinoma Previously Treated With Chemotherapy
Brief Title: Study of Everolimus in Patients With Thymoma and Thymic Carcinoma Previously Treated With Chemotherapy
Acronym: ONC-2010-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, principal Investigator, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2010-001
Record Dates: First submitted 2013-05-27; First posted 2014-01-29 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Thymoma and Thymic Carcinoma
Keywords: thymoma thymic carcinoma
MeSH Terms: conditions — Thymoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): oral everolimus
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus will be orally administered at the dosage of 10 mg once daily. Each cycle will be considered as 21 days of treatment. Tumor assessment will be done every two cycles.Treatment should be administered until documented disease progression, unacceptable toxicity, or patient refusal.
  Other Names: Afinitor

SUMMARY:
Given the high expression of IGF-1R and pAKT proteins in thymoma tissues, able to sensitize tumors to mTOR inhibition, and the anticancer activity of the mTOR inhibitors, clinical evaluation in thymoma and thymic carcinoma seems to be very interesting.

Patients will receive continuous treatment with oral everolimus 10 mg once daily.

Efficacy and safety profile of Everolimus will be evaluated.

DETAILED DESCRIPTION:
Patients will receive continuous treatment with oral everolimus 10 mg once daily. Study drug will be self-administered orally (two 5 mg tablets) daily in a fasting state or with a light fat-free meal. Each cycle will be considered as 21 days of treatment; safety was assessed every 21 days. Tumor assessement will be done every two cycles. Treatment should be administered until documented disease progression, unacceptable toxicity, or patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of invasive recurrent or metastatic thymoma or thymic carcinoma confirmed by pathologist.
* At least one prior platinum-containing chemotherapy regimen. There is no limit to the number of prior chemotherapy regimens received. Progressive disease should have been documented before entry into the study.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than 20 mm with conventional techniques or as greater than 10 mm with spiral CT scan.
* Patients must have recovered from toxicity related to prior therapy to at least to grade 1 (defined by CTCAE 3.0).
* No major surgery, radiation therapy, chemotherapy, biologic therapy (including any investigational agents), or hormonal therapy (other than replacement), within 4 weeks prior to entering the study.
* Life expectancy of at least 3 months.
* Performance status (ECOG)<=2
* Negative pregnancy test (if female in reproductive years)
* Adequate organ and marrow function (as defined below)
* Leukocytes >=3,000/mm, Absolute neutrophil count >=1,500/mm, Hemoglobin>= 9 g/dL, Platelets>= 100,000/mm, Total bilirubin >= 1.5 x institutional upper limit of normal (ULN), AST(SGOT)/ALT(SGPT)>= 3 x institutional ULN (5x if LFT elevations due to liver metastases, )Creatinine <= 1.5 x institutional ULN

Exclusion Criteria:

* Patients with symptomatic brain metastases. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 3 months without steroids may be enrolled at the discretion of the investigator.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to treatment
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Pregnant or breast feeding women
* Previous (within the last 5 years) or current malignancies at other sites, except for adequately treated basal cell or squamous cell skin cancer or in situ carcinoma of the cervix uteri
* Current enrollment in or participation in another therapeutic clinical trial within 4 weeks preceding treatment start.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgement of the Investigator, would make the patient inappropriate for entry into this study or could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
disease control rate | 6 months
  disease control rate (DCR), considered as complete response (CR) plus partial response (PR) plus stable disease (SD), of Everolimus monotherapy

SECONDARY OUTCOMES:
PFS | 6 months
  Progression free survival (PFS) will be evaluated from the date of treatment start until the date of progression or death whichever occurs first, otherwise until the last visit date.
Duration of Response | 6 months
  This endpoint is assessed in patients whose best tumor response is CR or PR as the time from the date of the first documentation of confirmed objective tumor response to the date of first documentation of objective tumor progression, objective tumor recurrence, or of death due progressive disease, whichever comes first
OS | 6 months
  Overall Survival (OS) will be evaluated from the date of treatment start until the date of death or last contact for patients alive at the end of the study.
FDG-PET imaging relations | 6 weeks
  To correlate response to therapy with changes in FDG-PET imaging at baseline and first restaging.
safety profile | 6 months
  Overall safety profile, evaluated on the basis of laboratory and clinical safety parameters
biomarkers expression | 6 months
  To perform immunohistochemistry for IGF-1R, pAKT ,mTOR, p-S6K, p-S6, p-4E-BP1, and pTEN expression in all pre-treatment tissue specimens of thymoma and thymic carcinoma and correlate with response and survival (PFS and OS).

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No
not planned

REFERENCES:
- [Derived] Zucali PA, De Pas T, Palmieri G, Favaretto A, Chella A, Tiseo M, Caruso M, Simonelli M, Perrino M, De Vincenzo F, Toffalorio F, Damiano V, Pasello G, Garbella E, Ali M, Conforti F, Ottaviano M, Cioffi A, De Placido S, Giordano L, Bertossi M, Destro A, Di Tommaso L, Santoro A. Phase II Study of Everolimus in Patients With Thymoma and Thymic Carcinoma Previously Treated With Cisplatin-Based Chemotherapy. J Clin Oncol. 2018 Feb 1;36(4):342-349. doi: 10.1200/JCO.2017.74.4078. Epub 2017 Dec 14. PMID 29240542